CLINICAL TRIAL: NCT00392756
Title: Role of Gonadotropin Pulsations in the Reversal of Hypogonadotropic Hypogonadism
Brief Title: Examination of Idiopathic Hypogonadotropic Hypogonadism (IHH)and Kallmann Syndrome (KS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, Harvard Reproductive Endocrine Sciences Center, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: U54HD028138-024; 5U54HD028138 (NIH)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Kallmann Syndrome; Hypogonadotropic Hypogonadism; GnRH Deficiency
Keywords: Kallmann Syndrome; Hypogonadotropic Hypogonadism; GnRH deficiency; Pulsatile GnRH
MeSH Terms: conditions — Kallmann Syndrome; Hypogonadism | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- off treatment (No Intervention): Subjects undergo the baseline evaluation off treatment
- GnRH Treatment (Experimental): Subjects receive long term pulsatile GnRH therapy
  Interventions: Drug: gonadotropin releasing hormone (GnRH)

INTERVENTIONS:
Drug: gonadotropin releasing hormone (GnRH) — pulsatile GnRH is delivered to adult men (18+ yrs) via portable microinfusion pump. A small dose (30 microliters) is delivered subcutaneously every 120 minutes. The initial dose is 25 ng/Kg which is increased until normal serum testosterone levels are achieved.
  Arms: GnRH Treatment

SUMMARY:
The purpose of the study is to examine how Kallmann syndrome (KS) and idiopathic hypogonadotropic hypogonadism (IHH) affect reproductive hormones. These disorders are caused by a defect in Gonadotropin Releasing Hormone (GnRH) secretion. GnRH is a hormone released by a small gland in the brain called the hypothalamus. When GnRH is released, it signals another gland in the brain, the pituitary, to secrete the reproductive hormones that influence sex hormone (testosterone, estrogen) levels and gamete (sperm, egg cell) production.

This study involves a detailed evaluation and 24-48 hours stay at the hospital.

In this study, males and females ages 16 and older with IHH have a detailed evaluation which involves an overnight study at the hospital. Some men (18 years and older) may continue on to receive treatment with pulsatile GnRH. This treatment replaces the hormone which is absent in IHH and results in normalized testosterone and typically is effective in developing fertility.

DETAILED DESCRIPTION:
The specific aims of this study are:

* To identify men and women with hypogonadotropic hypogonadism and to define the spectrum of abnormalities in GnRH secretion in these patients.
* To study the physiology and control of the reproductive system in the human male and female.
* To determine the relationship between glucose metabolism and testosterone levels in men with hypogonadotropic hypogonadism.
* To characterize the neuroendocrine and metabolic phenotype of participants with IHH and use this information to make genotype-phenotype correlations.

Despite variability in the triggers, timing, and pace of sexual maturity between species, all species utilize the final pathway of hypothalamic secretion of GnRH to initiate and maintain the reproductive axis. Thus, GnRH is required for reproductive competence in the human. The classic studies of Knobil and his colleagues in the 1970s clearly demonstrated that pulsatile release of GnRH from the hypothalamus is a prerequisite for physiologic gonadotrope function, with continuous stimulation resulting in a paradoxical decrease in gonadotrope responsiveness.

Absence, decreased frequency or decreased amplitude of pulsatile GnRH release results in the clinical syndrome of hypogonadotropic hypogonadism (HH). Deficient GnRH secretion may occur in isolation (idiopathic hypogonadotropic hypogonadism [IHH]), in association with anosmia (Kallmann syndrome [KS]) or as a result of a variety of structural and functional lesions of the hypothalamic-pituitary axis. The phenotypic expression of GnRH deficiency in the human demonstrates considerable heterogeneity, suggesting that patients with IHH and KS may represent part of a spectrum of isolated GnRH deficiency as opposed to representing discrete diagnostic subsets.

Defining the physiology of GnRH is critical to understanding the clinical heterogeneity of isolated GnRH deficiency. This protocol will utilize the disease model of HH to increase our understanding of the physiology of GnRH secretion. Examining the baseline characteristics of patients with isolated GnRH deficiency allows the determination of the normal requirements for endogenous GnRH secretion in the human.

Recent studies have revealed an association between hyperinsulinemia and low testosterone levels in men. This finding has been demonstrated in normal physiological conditions as well as in insulin resistant states. However, the causal nature and directionality of this relationship is not yet understood. Specifically, do lower testosterone levels cause insulin resistance resulting in hyperinsulinemia or vice versa? Because insulin resistance is an important risk factor for cardiovascular disease as well as type 2 diabetes, it is important to investigate this relationship for the implications it may have for prevention of and therapeutic interventions for these disorders.

ELIGIBILITY:
Eligibility

Ages Eligible for Study:

* Adolescents (16-17yrs)
* Adults (18 years and older)

  * Genders Eligible for Study:
* Male and Female

  * Accepts Healthy Volunteers:
* No

Criteria

Inclusion Criteria:

* adolescent boys (age 16-17 years) and adult male individuals (age 18 years and older) with a single serum sample demonstrating low testosterone in association with low or inappropriately normal gonadotropin levels
* adolescent girls (age 16-17 years) and adult female individuals (age 18 years and older) with a single serum sample demonstrating low estradiol (estrogen) in association with low or inappropriately normal gonadotropin levels
* suitable male and female hypogonadotropic hypogonadal subjects

Exclusion Criteria:

* no specific exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 1989-04; Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
endogenous LH secretion pattern | 8 to 24 hours

SECONDARY OUTCOMES:
testicular volume | up to 2 years
sperm count | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Belchetz PE, Plant TM, Nakai Y, Keogh EJ, Knobil E. Hypophysial responses to continuous and intermittent delivery of hypopthalamic gonadotropin-releasing hormone. Science. 1978 Nov 10;202(4368):631-3. doi: 10.1126/science.100883.
- [Background] Seminara SB, Hayes FJ, Crowley WF Jr. Gonadotropin-releasing hormone deficiency in the human (idiopathic hypogonadotropic hypogonadism and Kallmann's syndrome): pathophysiological and genetic considerations. Endocr Rev. 1998 Oct;19(5):521-39. doi: 10.1210/edrv.19.5.0344. No abstract available. PMID 9793755
- [Background] Arimura A, Kastin AJ, Gonzalez-Barcena D, Siller J, Weaver RE, Schally AV. Disappearance of LH-releasing hormone in man as determined by radioimmunoassay. Clin Endocrinol (Oxf). 1974 Oct;3(4):421-5. doi: 10.1111/j.1365-2265.1974.tb02812.x. No abstract available. PMID 4609640
- [Background] Pimstone B, Epstein S, Hamilton SM, LeRoith D, Hendricks S. Metabolic clearance and plasma half disappearance time of exogenous gonadotropin releasing hormone in normal subjects and in patients with liver disease and chronic renal failure. J Clin Endocrinol Metab. 1977 Feb;44(2):356-60. doi: 10.1210/jcem-44-2-356. PMID 320223
- [Background] Clarke IJ, Cummins JT. The temporal relationship between gonadotropin releasing hormone (GnRH) and luteinizing hormone (LH) secretion in ovariectomized ewes. Endocrinology. 1982 Nov;111(5):1737-9. doi: 10.1210/endo-111-5-1737. No abstract available. PMID 6751801
- [Background] Karsch FJ, Bowen JM, Caraty A, Evans NP, Moenter SM. Gonadotropin-releasing hormone requirements for ovulation. Biol Reprod. 1997 Feb;56(2):303-9. doi: 10.1095/biolreprod56.2.303. PMID 9116125
- [Background] Spratt DI, O'Dea LS, Schoenfeld D, Butler J, Rao PN, Crowley WF Jr. Neuroendocrine-gonadal axis in men: frequent sampling of LH, FSH, and testosterone. Am J Physiol. 1988 May;254(5 Pt 1):E658-66. doi: 10.1152/ajpendo.1988.254.5.E658. PMID 3129947
- [Background] Hayes FJ, McNicholl DJ, Schoenfeld D, Marsh EE, Hall JE. Free alpha-subunit is superior to luteinizing hormone as a marker of gonadotropin-releasing hormone despite desensitization at fast pulse frequencies. J Clin Endocrinol Metab. 1999 Mar;84(3):1028-36. doi: 10.1210/jcem.84.3.5579. PMID 10084591
- [Background] Whitcomb RW, Crowley WF Jr. Clinical review 4: Diagnosis and treatment of isolated gonadotropin-releasing hormone deficiency in men. J Clin Endocrinol Metab. 1990 Jan;70(1):3-7. doi: 10.1210/jcem-70-1-3. No abstract available. PMID 2403572
- [Background] Simon D, Preziosi P, Barrett-Connor E, Roger M, Saint-Paul M, Nahoul K, Papoz L. Interrelation between plasma testosterone and plasma insulin in healthy adult men: the Telecom Study. Diabetologia. 1992 Feb;35(2):173-7. doi: 10.1007/BF00402551. PMID 1547923
- [Background] Lichtenstein MJ, Yarnell JW, Elwood PC, Beswick AD, Sweetnam PM, Marks V, Teale D, Riad-Fahmy D. Sex hormones, insulin, lipids, and prevalent ischemic heart disease. Am J Epidemiol. 1987 Oct;126(4):647-57. doi: 10.1093/oxfordjournals.aje.a114704. PMID 3307391
- [Background] Seidell JC, Bjorntorp P, Sjostrom L, Kvist H, Sannerstedt R. Visceral fat accumulation in men is positively associated with insulin, glucose, and C-peptide levels, but negatively with testosterone levels. Metabolism. 1990 Sep;39(9):897-901. doi: 10.1016/0026-0495(90)90297-p. PMID 2202881
- [Background] Pasquali R, Casimirri F, Cantobelli S, Melchionda N, Morselli Labate AM, Fabbri R, Capelli M, Bortoluzzi L. Effect of obesity and body fat distribution on sex hormones and insulin in men. Metabolism. 1991 Jan;40(1):101-4. doi: 10.1016/0026-0495(91)90199-7. PMID 1984562
- [Background] Barrett-Connor E. Lower endogenous androgen levels and dyslipidemia in men with non-insulin-dependent diabetes mellitus. Ann Intern Med. 1992 Nov 15;117(10):807-11. doi: 10.7326/0003-4819-117-10-807. PMID 1416554
- [Background] Andersson B, Marin P, Lissner L, Vermeulen A, Bjorntorp P. Testosterone concentrations in women and men with NIDDM. Diabetes Care. 1994 May;17(5):405-11. doi: 10.2337/diacare.17.5.405. PMID 8062607
- [Background] Ducimetiere P, Eschwege E, Papoz L, Richard JL, Claude JR, Rosselin G. Relationship of plasma insulin levels to the incidence of myocardial infarction and coronary heart disease mortality in a middle-aged population. Diabetologia. 1980 Sep;19(3):205-10. doi: 10.1007/BF00275270. PMID 6997122
- [Background] Filippi G. Klinefelter's syndrome in Sardinia. Clinical report of 265 hypogonadic males detected at the time of military check-up. Clin Genet. 1986 Oct;30(4):276-84. PMID 3791676
- [Background] Fromantin M, Gineste J, Didier A, Rouvier J. [Impuberism and hypogonadism at induction into military service. Statistical study]. Probl Actuels Endocrinol Nutr. 1973 May 3;16:179-99. No abstract available. French. PMID 4147392
- [Background] Filicori M, Butler JP, Crowley WF Jr. Neuroendocrine regulation of the corpus luteum in the human. Evidence for pulsatile progesterone secretion. J Clin Invest. 1984 Jun;73(6):1638-47. doi: 10.1172/JCI111370. PMID 6427277
- [Background] Narasimha Rao P, Moore PH Jr. Synthesis of new steroid haptens for radioimmunoassay. Part I. 15beta-Carboxyethylmercaptotestosterone-bovine serum albumin conjugate. Measurement of testosterone in male plasma without chromatography. Steroids. 1976 Jul;28(1):101-9. doi: 10.1016/0039-128x(76)90129-x. PMID 960143
- [Background] Groome NP, Illingworth PJ, O'Brien M, Pai R, Rodger FE, Mather JP, McNeilly AS. Measurement of dimeric inhibin B throughout the human menstrual cycle. J Clin Endocrinol Metab. 1996 Apr;81(4):1401-5. doi: 10.1210/jcem.81.4.8636341.
- [Background] Landy H, Schneyer AL, Whitcomb RW, Crowley WF Jr. Validation of highly specific and sensitive radioimmunoassays for lutropin, follitropin, and free alpha subunit in unextracted urine. Clin Chem. 1990 Feb;36(2):340-4. PMID 2105862
- [Background] Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Diabetes Care. 1997 Jul;20(7):1183-97. doi: 10.2337/diacare.20.7.1183. No abstract available. PMID 9203460
- [Result] Pitteloud N, Hayes FJ, Dwyer A, Boepple PA, Lee H, Crowley WF Jr. Predictors of outcome of long-term GnRH therapy in men with idiopathic hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2002 Sep;87(9):4128-36. doi: 10.1210/jc.2002-020518. PMID 12213860
- [Result] Hayes FJ, Seminara SB, Crowley WF Jr. Hypogonadotropic hypogonadism. Endocrinol Metab Clin North Am. 1998 Dec;27(4):739-63, vii. doi: 10.1016/s0889-8529(05)70039-6. PMID 9922906
- [Result] Nachtigall LB, Boepple PA, Pralong FP, Crowley WF Jr. Adult-onset idiopathic hypogonadotropic hypogonadism--a treatable form of male infertility. N Engl J Med. 1997 Feb 6;336(6):410-5. doi: 10.1056/NEJM199702063360604. PMID 9010147
- [Result] Whitcomb RW, Crowley WF Jr. Hypogonadotropic hypogonadism: gonadotropin-releasing hormone therapy. Curr Ther Endocrinol Metab. 1997;6:353-5. No abstract available. PMID 9174769
- [Result] Crowley WF, Whitcomb RW. Gonadotropin-releasing hormone deficiency in men: diagnosis and treatment with exogenous gonadotropin-releasing hormone. Am J Obstet Gynecol. 1990 Nov;163(5 Pt 2):1752-8. doi: 10.1016/0002-9378(90)91440-n. PMID 2122732
- [Result] Finkelstein JS, Spratt DI, O'Dea LS, Whitcomb RW, Klibanski A, Schoenfeld DA, Crowley WF Jr. Pulsatile gonadotropin secretion after discontinuation of long term gonadotropin-releasing hormone (GnRH) administration in a subset of GnRH-deficient men. J Clin Endocrinol Metab. 1989 Aug;69(2):377-85. doi: 10.1210/jcem-69-2-377. PMID 2502554
- [Result] Spratt DI, Carr DB, Merriam GR, Scully RE, Rao PN, Crowley WF Jr. The spectrum of abnormal patterns of gonadotropin-releasing hormone secretion in men with idiopathic hypogonadotropic hypogonadism: clinical and laboratory correlations. J Clin Endocrinol Metab. 1987 Feb;64(2):283-91. doi: 10.1210/jcem-64-2-283. PMID 3098771
- [Result] Spratt DI, Finkelstein JS, O'Dea LS, Badger TM, Rao PN, Campbell JD, Crowley WF Jr. Long-term administration of gonadotropin-releasing hormone in men with idiopathic hypogonadotropic hypogonadism. A model for studies of the hormone's physiologic effects. Ann Intern Med. 1986 Dec;105(6):848-55. doi: 10.7326/0003-4819-105-6-848. PMID 3096182
- [Result] Spratt DI, Crowley WF Jr, Butler JP, Hoffman AR, Conn PM, Badger TM. Pituitary luteinizing hormone responses to intravenous and subcutaneous administration of gonadotropin-releasing hormone in men. J Clin Endocrinol Metab. 1985 Nov;61(5):890-5. doi: 10.1210/jcem-61-5-890. PMID 3900124
- [Result] Hoffman AR, Crowley WF Jr. Induction of puberty in men by long-term pulsatile administration of low-dose gonadotropin-releasing hormone. N Engl J Med. 1982 Nov 11;307(20):1237-41. doi: 10.1056/NEJM198211113072003. PMID 6813732
- [Result] Crowley WF Jr, Beitins IZ, Vale W, Kliman B, Rivier J, Rivier C, McArthur JW. The biologic activity of a potent analogue of gonadotropin-releasing hormone in normal and hypogonadotropic men. N Engl J Med. 1980 May 8;302(19):1052-7. doi: 10.1056/NEJM198005083021903. PMID 6767977
- [Result] Raivio T, Falardeau J, Dwyer A, Quinton R, Hayes FJ, Hughes VA, Cole LW, Pearce SH, Lee H, Boepple P, Crowley WF Jr, Pitteloud N. Reversal of idiopathic hypogonadotropic hypogonadism. N Engl J Med. 2007 Aug 30;357(9):863-73. doi: 10.1056/NEJMoa066494. PMID 17761590
- [Result] Pitteloud N, Hayes FJ, Boepple PA, DeCruz S, Seminara SB, MacLaughlin DT, Crowley WF Jr. The role of prior pubertal development, biochemical markers of testicular maturation, and genetics in elucidating the phenotypic heterogeneity of idiopathic hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2002 Jan;87(1):152-60. doi: 10.1210/jcem.87.1.8131. PMID 11788640
- [Result] Shaw ND, Seminara SB, Welt CK, Au MG, Plummer L, Hughes VA, Dwyer AA, Martin KA, Quinton R, Mericq V, Merino PM, Gusella JF, Crowley WF Jr, Pitteloud N, Hall JE. Expanding the phenotype and genotype of female GnRH deficiency. J Clin Endocrinol Metab. 2011 Mar;96(3):E566-76. doi: 10.1210/jc.2010-2292. Epub 2011 Jan 5. PMID 21209029
- [Derived] Delaney A, Volochayev R, Meader B, Lee J, Almpani K, Noukelak GY, Henkind J, Chalmers L, Law JR, Williamson KA, Jacobsen CM, Buitrago TP, Perez O, Cho CH, Kaindl A, Rauch A, Steindl K, Garcia JE, Russell BE, Prasad R, Mondal UK, Reigstad HM, Clements S, Kim S, Inoue K, Arora G, Salnikov KB, DiOrio NP, Prada R, Capri Y, Morioka K, Mizota M, Zechi-Ceide RM, Kokitsu-Nakata NM, Tonello C, Vendramini-Pittoli S, da Silva Dalben G, Balasubramanian R, Dwyer AA, Seminara SB, Crowley WF, Plummer L, Hall JE, Graham JM, Lin AE, Shaw ND. Insight Into the Ontogeny of GnRH Neurons From Patients Born Without a Nose. J Clin Endocrinol Metab. 2020 May 1;105(5):1538-51. doi: 10.1210/clinem/dgaa065. PMID 32034419